CLINICAL TRIAL: NCT04775563
Title: COVID-19 Vaccine Hesitancy Among Mexican Rheumatic Diseases Patients
Brief Title: COVID-19 Vaccine Hesitancy Among Rheumatic Diseases Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, PI, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE-3639
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: vaccines, rheumatic diseases
MeSH Terms: conditions — COVID-19; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatic diseases outpatients: All the rheumatic diseases outpatients from the National Institute of Medical Sciences and General Hospital.
  Interventions: Other: COVID-19 vaccine hesitancy scale in rheumatic diseases; Other: COVID-19 vaccine hesitancy associated factors

INTERVENTIONS:
Other: COVID-19 vaccine hesitancy scale in rheumatic diseases — The instrument was developed by Freeman et al, prior to its application, translation, cultural adaptation, and validation were performed.
Other: COVID-19 vaccine hesitancy associated factors — The instrument includes questions about the doctor-patient relationship, perception of the COVID-19 vaccine, perception of risk of COVID-19 infection, perception of the severity of the pandemic in Mexico, perception of the severity of their rheumatic disease, perception of the control of comorbidities, perception of the intensity of the immunosuppressive treatment, positioning of the patient towards vaccines for COVID-19

SUMMARY:
Rheumatological diseases (RD) are an important group of different clinical entities and specific diseases that affect a significant proportion of the world population. In Mexico, the RD have a relevant representation in the adult population. COVID-19 vaccination has been proposed as a measure to contain the COVID-19 pandemic. The vaccines have been shown to be effective and reasonably safe in the population without significant risk factors, which has allowed their approval to attend the health emergency. At present, there is little scientific information that allows a solid recommendation on vaccination for COVID-19 in patients with RD, although most authorities have spoken in favor of vaccination in immunocompromised patients, as are a relevant number of patients with RD. However, it is desirable to achieve herd immunity to facilitate the impact of vaccination on the transmission of SARS-CoV-2 infection. For this, it is required that around 70% -80% of the target population be vaccinated, which implies not only access to the vaccine but also accepting to be vaccinated.

Vaccine hesitancy is defined as the delay or refusal to accept the vaccine when it is available by health services. Sometimes, they conceptualize it as a continuum and also includes the high demand from the population for the vaccine; In this continuum, there are variations in acceptance and rejection and multiple possible combinations, from acceptance with great concern about the decision to rejection of certain vaccines but not others. It is a complex, contextual, changing phenomenon, specific for each vaccine and the referred disease and probably influenced by cultural determinants.

DETAILED DESCRIPTION:
The objectives are:

1. - To measure the phenomenon of vaccine hesitancy in Mexican patients with RD from two Health Institutions in Mexico City.
2. - Translate and adapt the "Oxford Covid-19 vaccine hesitancy scale" to patients with RD and validate this version in a population of patients with RD from two Health Institutions in Mexico City
3. Explore factors associated with the phenomenon of vaccine hesitancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a rheumatic disease diagnosis according to their primary rheumatologist who agree to participate

Exclusion Criteria:

* Patients with a not confirmed rheumatic disease

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the rheumatic diseases outpatients from the National Institute of Medical Sciences and Nutrition and General Hospital.
Sampling Method: Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Measure the phenomenon of vaccine hesitancy among rheumatic diseases patients | At study inclusion
  Identify the percentage of patients with rheumatic diseases that present COVID-19 vaccine hesitancy using the instrument developed by Freeman et al (translation, cultural adaptation, and validation performed)

SECONDARY OUTCOMES:
Identify factors associated with COVID-19 vaccine hesitancy among rheumatic diseases patients | At study inclusion
  Identify factors associated with COVID-19 vaccine hesitancy among rheumatic diseases patients using an instrument locally development

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No